CLINICAL TRIAL: NCT04727970
Title: A Phase I Open-Label Pilot Study to Investigate the Feasibility, Safety, Tolerability and Efficacy of Daily Administration of Tricaprilin in Subjects with Infantile Spasms
Brief Title: Tricaprilin Infantile Spasms Pilot Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cerecin (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC-21-024
Record Dates: First submitted 2021-01-19; First posted 2021-01-27 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Infantile Spasm
MeSH Terms: conditions — Spasms, Infantile | interventions — tricaprylin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tricaprilin (Experimental): Tricaprilin will be administered for 5-21 days. The total daily dose (individual per subject up to a maximum of 10g/kg/day) will be split into 4 doses administered orally, approximately every 6 hours.
  Interventions: Drug: Tricaprilin

INTERVENTIONS:
Drug: Tricaprilin — Tricaprilin will be emulsified in infant formula/milk
  Other Names: AC-OL-01

SUMMARY:
The purpose of this study is to assess the safety, tolerability, and efficacy of tricaprilin in subjects with infantile spasms. This is a single-arm, open-label, pilot study in up to 10 subjects with infantile spasms.

Upon completion of the main phase, subjects who exhibit improvement in seizure control and who tolerate the compound will be offered continued use of the IMP until benefit-risk ratio is no longer favourable, in a one-year open-label extension phase, available to Australian participants only.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female infants ages 3 months to 24 months, inclusive, at the time of parent/legal guardian signing the informed consent
2. Clinical diagnosis of IS, confirmed by analysis of a 24-hour video-electroencephalogram (vEEG) recording, including at least one documented spasm
3. Continued infantile spasms despite adequate treatment with oral prednisolone (or adrenocorticotropic hormone [ACTH]) and vigabatrin
4. If being treated with concomitant ASDs (other than ketogenic therapies/diet), current ASDs have been at a constant daily dose for at least 1 week.
5. Subject is taking no more than 3 concomitant ASDs

Exclusion Criteria:

1. Subject considered by the Investigator, for any reason, to be an unsuitable candidate to receive the investigational product
2. Significant and active pre-existing cardiovascular, renal, liver, infectious, or other systemic disease
3. Subject has clinically significant renal impairment
4. Clinically significant abnormality on ECG that, in the opinion of the Investigator, increases the safety risks of participating in the study
5. Known or suspected allergy to the investigational product
6. Known history of aspiration pneumonia within the past year
7. Previous participation in another clinical study of the investigational product or received any investigational drug, device, or therapy within 30 days of study entry or within five half-lives of another investigational drug
8. Within 14 days of screening, subject has:

   1. received therapy with felbamate, cannabinoids, ketogenic diet, or vagus nerve stimulation
   2. received therapy with ACTH, prednisolone or other steroid
9. Pre-existing lethal or potentially lethal condition other than infantile spasms
10. Previous failure to respond to an appropriate trial (at least 2 weeks) of the ketogenic diet

Ages: 3 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-12-04 (Actual); Study Completion 2023-12-04 (Actual)

PRIMARY OUTCOMES:
To determine the safety of daily administration of tricaprilin in subjects with Infantile Spasms (IS) | Up to end of study (Day 5 to 21; depending on subject)
  Treatment emergent adverse events
To determine the safety and tolerability of daily administration of tricaprilin in subjects with Infantile Spasms (IS) | Up to end of study (Day 5 to 21; depending on subject)
  Brussels Infant and Toddler Stool Scale; the scale consists of 4 categories: hard, formed, loose or watery. The category of stools per subject will be compared between baseline and during the study.
Extension Phase (for Australian sites only): To determine the safety of daily long-term administration of tricaprilin in subjects with Infantile Spasms (IS) | End of main phase treatment period to end of extension phase (1-year period)
  Treatment emergent adverse events

SECONDARY OUTCOMES:
Change in spasm frequency based on caregiver spasm/seizure diary | Baseline (1-week period) to end of treatment period (1-week period)
  Number of clusters and mean cluster duration
Change in spasm frequency based on 24-hour video-EEG | Baseline (1-week period) to end of treatment period (1-week period)
  Number of clusters and mean cluster duration
Extension Phase (for Australian sites only): Change in spasm frequency based on caregiver spasm/seizure diary | End of main phase treatment period to end of extension phase (1-year period)
  Number of clusters and mean cluster duration

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Cerecin
Locations (4):
- Australia (3):
  - Sydney Children's Hospital, Randwick, New South Wales
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Royal Children's Hospital Melbourne, Parkville, Victoria
- KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No